CLINICAL TRIAL: NCT07329413
Title: Does Anterior Disc Displacement With Reduction Affect Postoperative Pain After Root Canal Treatment in Patients With Symptomatic Apical Periodontitis? A Prospective, Quasi-Experimental Controlled Study
Brief Title: Effect of Anterior Disc Displacement With Reduction on Postoperative Pain After Root Canal Treatment
Acronym: TMD-POSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, burcu revi, Principal Investigator, Recep Tayyip Erdogan University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/82; 2025/82 (Other: Recep Tayyip Erdoğan University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Apical Periodontitis; Temporomandibular Disorders (TMDs); Anterior Disc Displacement
Keywords: Endodontics; Postoperative pain; Root Canal Therapy; Temporomandibular Joint; Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups based on the presence or absence of anterior disc displacement with reduction. Both groups received root canal treatment using the same standardized clinical protocol, and outcomes were evaluated in parallel.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An oral diagnosis and radiology specialist with more than 10 years of clinical experience evaluated the patients' endodontic treatment needs and performed the temporomandibular joint examination. Patients diagnosed with anterior disc displacement with reduction according to the Diagnostic Criteria for Temporomandibular Disorders were assigned to the experimental group, while individuals without temporomandibular joint disorders constituted the control group.
  At this stage, both the participants and the clinician performing the root canal treatments were blinded to the temporomandibular joint status of the patients (double-blind). Group allocation was concealed until completion of the data analysis, resulting in a triple-blind study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADDR group (Experimental): Patients diagnosed with anterior disc displacement with reduction according to the Diagnostic Criteria for Temporomandibular Disorders.
  Interventions: Procedure: Single-Visit Conventional Root Canal Treatment Using Nickel-Titanium Rotary Instruments (Endoart Smart Gold); Drug: Ibuprofen 400 mg (if necessary)
- Control group (Active Comparator): Patients without any temporomandibular joint pathology.
  Interventions: Procedure: Single-Visit Conventional Root Canal Treatment Using Nickel-Titanium Rotary Instruments (Endoart Smart Gold); Drug: Ibuprofen 400 mg (if necessary)

INTERVENTIONS:
Procedure: Single-Visit Conventional Root Canal Treatment Using Nickel-Titanium Rotary Instruments (Endoart Smart Gold) — All endodontic treatments were performed in a single visit by a single operator (BR) with six years of clinical experience, using a standardized treatment protocol. Only one tooth per patient was included in the study. Inferior alveolar nerve block anesthesia was administered. After rubber dam isolation, access cavities were prepared. Working length was determined using an electronic apex locator set at 0.5 mm short of the apical foramen and confirmed with periapical radiography. Root canals were prepared using Endoart Smart Gold rotary instruments (Inci Dental, Istanbul, Türkiye) up to size 25/.04 for mesial canals and 30/.04 for distal canals. If insufficient apical instrumentation was detected, canal enlargement was extended up to a maximum of two sizes larger, according to canal length and anatomy. Following canal preparation, final irrigation was performed. The canals were obturated using the lateral condensation technique with a resin-based root canal sealer.
Drug: Ibuprofen 400 mg (if necessary) — Ibuprofen (oral analgesic) was prescribed to all patients who underwent root canal treatment and was recommended for use only in case of postoperative pain.

SUMMARY:
The aim of this study is to evaluate the impact of anterior disc displacement with reduction (ADDR) on postoperative pain following root canal treatment in patients diagnosed with symptomatic apical periodontitis.

DETAILED DESCRIPTION:
This prospective clinical study included individuals diagnosed with symptomatic apical periodontitis who had a vital mandibular molar tooth and were diagnosed with anterior disc displacement with reduction (ADDR) according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) (n = 45), as well as individuals without any temporomandibular joint pathology (n = 45). Following patient dropouts, a total of 70 patients with complete and eligible data were included in the final analysis, with 35 participants in each group.

All root canal treatments were performed by the same clinician using a standardized treatment protocol. Postoperative pain intensity was assessed using the Numeric Rating Scale at 6 and 12 hours and at 1, 2, 3, 5, and 7 days after treatment. In addition, joint sounds, joint pain, and maximum mouth opening were recorded in the preoperative period and at the 7-day postoperative follow-up, and their associations with postoperative pain were analyzed.

The findings of this study provide insight into the relationship between temporomandibular joint disorders and endodontic postoperative pain and may contribute to improved clinical understanding.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65 years with no systemic disease
* Patients diagnosed with symptomatic apical periodontitis
* Presence of a vital permanent mandibular first or second molar tooth requiring root canal treatment
* Teeth with no radiographic evidence of periapical changes or only slight widening of the periodontal ligament space
* Patients reporting preoperative spontaneous pain with a Numeric Rating Scale (NRS) score between 4 and 10 (moderate pain: 4-6; severe pain: 7-10)
* Patients reporting pain intensity of 4 or higher on the NRS during percussion testing
* Patients diagnosed with isolated anterior disc displacement with reduction according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) (experimental group) or patients without any temporomandibular joint disorder or pathology (control group)

Exclusion Criteria:

* Teeth found to have necrotic pulp tissue during access cavity preparation
* Patients in whom the study tooth was not located on the same side as the temporomandibular joint diagnosed with anterior disc displacement with reduction
* Occurrence of any endodontic complications during treatment
* Use of medications that could affect pain perception (e.g., analgesics or anti-inflammatory drugs) within at least 12 hours before treatment, or use of systemic antibiotics within one month prior to enrollment
* History of major jaw trauma, dentofacial deformities, or previous temporomandibular joint surgery
* Concurrent use of steroids, muscle relaxants, or narcotic medications
* History of diagnosed neuropathic pain, myofascial pain, neuralgic pain, or chronic headache disorders
* Presence of periodontal disease (probing depth > 5 mm or tooth mobility greater than Grade I) or teeth lacking adequate coronal structure
* Teeth without occlusal contact or with premature contacts, patients with bruxism or clenching habits, or patients with fewer than three teeth on one side of the mandible
* Inability to read, understand, or complete the pain assessment scale or to provide the required follow-up data
* Presence of significant cognitive impairment (e.g., communication deficits, intellectual disability) or diagnosed psychiatric disorders (e.g., depression, anxiety disorders)
* Presence of immature teeth or teeth with open apices
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | 6, 12 hours 1, 2, 3, 5 and 7 days postoperatively
  To evaluate postoperative pain, each patient was provided with a pain diary after root canal treatment and was instructed to record pain intensity using the Numeric Rating Scale (NRS). Detailed instructions on how to use the NRS were given to all participants. Pain intensity was recorded at 6, 12, 24, 48, and 72 hours and at 5 and 7 days after treatment. Patients were prescribed 400 mg ibuprofen for use only in cases of severe pain. Data from patients who used analgesics during the follow-up period were excluded from the analysis.

SECONDARY OUTCOMES:
Maximum mouth opening | Baseline and 7 days postoperatively
  Maximum mouth opening was measured in millimeters using a digital caliper during the preoperative examination and at the 7-day postoperative follow-up.
Temporomandibular joint pain and percussion sensitivity | Baseline and 7 days postoperatively
  Temporomandibular joint pain and percussion sensitivity of the treated tooth were evaluated using the Numeric Rating Scale during the preoperative period and at the 7-day postoperative follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Edanur Maraş, DDS, PhD, Principal Investigator — Recep Tayyip Erdoğan University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.